CLINICAL TRIAL: NCT03651271
Title: An Exploratory Study of Nivolumab With or Without Ipilimumab According to the Percentage of Tumoral CD8 Cells in Participants With Advanced Metastatic Cancer
Brief Title: Nivolumab With or Without Ipilimumab in Advanced Metastatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Parker Institute for Cancer Immunotherapy (Other)
Collaborators: Bristol-Myers Squibb (Industry); Cancer Research Institute, New York City (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PICI0025
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Results first posted 2024-01-17 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Advanced Metastatic Cancer; Advanced Prostate Cancer
MeSH Terms: interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- "Hot" tumors for Advanced Metastatic Cancer (Experimental): Participants with ≥ 15% CD8 cells in their tumor biopsies (ie, CD8 high tumors) will be treated with single-agent nivolumab. At PD, participants will be allowed to add ipilimumab.
  Interventions: Biological: Nivolumab Monotherapy
- "Cold" tumors for Advanced Metastatic Cancer (Experimental): Participants with < 15% CD8 cells in their tumor biopsies (ie, CD8 low tumors) will be treated with nivolumab in combination with ipilimumab.
  Interventions: Biological: Nivolumab and Ipilimumab and Combination for Metastatic Cancer
- "Hot" tumors for Advanced Prostate Cancer (Experimental): Participants with ≥ 15% CD8 cells in their tumor biopsies (ie, CD8 high tumors) will be treated with single-agent nivolumab. At PD, participants will be allowed to add ipilimumab.
  Interventions: Biological: Nivolumab Monotherapy
- "Cold" tumors for Advanced Prostate Cancer Cohort A (Experimental): Participants with < 15% CD8 cells in their tumor biopsies (ie, CD8 low tumors) will be treated with nivolumab in combination with ipilimumab.
  Interventions: Biological: Nivolumab and Ipilimumab (3 mg/kg) Combination for Prostate Cancer
- "Cold" tumors for Advanced Prostate Cancer Cohort B (Experimental): Participants with < 15% CD8 cells in their tumor biopsies (ie, CD8 low tumors) will be treated with nivolumab in combination with ipilimumab.
  Interventions: Biological: Nivolumab and Ipilimumab (5 mg/kg) Combination for Prostate Cancer

INTERVENTIONS:
Biological: Nivolumab Monotherapy — Single-agent nivolumab will be administered at 360 mg IV Q3W. Participants who continue to show clinical benefit after the first disease assessment will receive nivolumab 480 mg IV Q4W until PD or intolerable toxicity.
  Arms: "Hot" tumors for Advanced Metastatic Cancer; "Hot" tumors for Advanced Prostate Cancer
Biological: Nivolumab and Ipilimumab and Combination for Metastatic Cancer — For nivolumab and ipilimumab combination therapy, nivolumab will be administered at 360 mg IV Q3W, and ipilimumab will be administered at 1 mg/kg IV Q3W for the first 2 doses and then Q6W for the 3rd and 4th doses, followed by single-agent nivolumab 480 mg IV Q4W until PD or intolerable toxicity.
  Arms: "Cold" tumors for Advanced Metastatic Cancer
Biological: Nivolumab and Ipilimumab (3 mg/kg) Combination for Prostate Cancer — For nivolumab and ipilimumab combination therapy, CD8 low arm, approximately 10 participants will be randomly allocated into 1 of 2 cohorts, using different doses of ipilimumab administered in 6-week cycles. Participants assigned to Prostate Cohort A will receive nivolumab 1 mg/kg Q3W and ipilimumab 3 mg/kg every 6 weeks (Q6W) for 2 cycles, then nivolumab maintenance 480 mg Q4W until PD or intolerable toxicity. If the safety profile of Prostate Cohort B is deemed unacceptable, an additional 10 participants will be enrolled in Prostate Cohort A.
  Arms: "Cold" tumors for Advanced Prostate Cancer Cohort A
Biological: Nivolumab and Ipilimumab (5 mg/kg) Combination for Prostate Cancer — For nivolumab and ipilimumab combination therapy, CD8 low arm, approximately 10 participants will be randomly allocated into 1 of 2 cohorts, using different doses of ipilimumab administered in 6-week cycles. Participants assigned to Prostate Cohort B will receive nivolumab 1 mg/kg Q3W and ipilimumab 5 mg/kg Q6W for 2 cycles, then nivolumab maintenance 480 mg Q4W until PD or intolerable toxicity. If Prostate Cohort B is determined to have a tolerable safety profile, an additional 10 participants will be enrolled to receive nivolumab 1 mg/kg Q3W and ipilimumab 5 mg/kg Q6W for 2 cycles, then nivolumab maintenance 480 mg Q4W until PD or intolerable toxicity.
  Arms: "Cold" tumors for Advanced Prostate Cancer Cohort B

SUMMARY:
This is an open-label, exploratory study to evaluate nivolumab with or without ipilimumab based on percentage of tumoral CD8 cells at the time of treatment in participants with varying advanced solid tumors. Participants who have a tumor with ≥ 15% CD8 cells (classified as CD8 high) will receive nivolumab monotherapy, and participants who have a tumor with < 15% CD8 cells (classified as CD8 low) will receive ipilimumab in combination with nivolumab.

DETAILED DESCRIPTION:
The aim of this study is to provide a prospective classification of CD8 high (immunologically "hot") versus CD8 low (immunologically "cold") tumors at the time of treatment, based on the percentage of CD8 cells in a tumor biopsy, and to address the predictive value of the CD8 biomarker for selecting patients for treatment with nivolumab with or without ipilimumab.

A total of up to approximately 200 participants with advanced metastatic cancer will be enrolled. Ongoing monitoring for safety and futility will be implemented based on the method of Thall and colleagues (Thall et al, 1995) separately in the CD8 high and CD8 low tumor groups. Single-agent nivolumab will be administered at 360 mg intravenously (IV) every 3 weeks (Q3W). Participants who continue to show clinical benefit after the first disease assessment will receive nivolumab 480 mg IV every 4 weeks (Q4W) until progressive disease (PD) or intolerable toxicity. At PD, participants will be allowed to add ipilimumab. For nivolumab and ipilimumab combination therapy, nivolumab will be administered at 360 mg IV Q3W, and ipilimumab will be administered at 1 mg/kg IV Q3W for the first 2 doses and then every 6 weeks for the 3rd and 4th doses, followed by nivolumab 480 mg IV Q4W until PD or intolerable toxicity. After receipt of the first dose of ipilimumab, the Investigator may determine (based on clinical symptoms) the number of future doses of ipilimumab the participant will receive, for a maximum of 4 doses. Participants who stop ipilimumab dosing early due to toxicities, may start nivolumab maintenance (ie, 4 doses [12 weeks] of nivolumab following the first dose).

Advanced prostate cancer participants with tumoral CD8 ≥ 15% will be enrolled in the nivolumab monotherapy arm. A total of approximately 20 participants with Advanced Prostate Cancer and tumoral CD8 < 15% will be allocated to 1 of 2 cohorts using combinations of ipilimumab and nivolumab.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥ 18 years of age inclusive, at the time of signing the informed consent.
2. Male or female participants of child-producing potential must agree to use contraception or avoidance of pregnancy measures during the study and for 7 and 5 months, respectively, after the last dose.
3. Females of childbearing potential must have a negative serum or urine pregnancy test.
4. Histologically or cytologically confirmed cancer that is metastatic, unresectable, or recurrent and are responsive to immunomodulation (ie, with US Prescribing Information [USPI]). Participants who have failed or refused available approved treatment options are eligible to participate.
5. Participants who have received prior immunotherapy, including prior anti-PD-1 or anti-PD-L1 therapies, will be allowed to participate in this study.

   1. Participants who received prior anti-PD-1 or anti-PD-L1 may participate only if their prior anti-PD-1 or anti-PD-L1 monotherapy or combination therapy were NOT the last treatment prior to participation on this study.
   2. Participants who had prior immunotherapies and experienced Grade 1-2 immune-related adverse event (irAE) must have documentation that their irAEs are ≤ Grade 1 or baseline using current Common Terminology Criteria for Adverse Events v5.0 (CTCAE v5.0) and participants must be off steroid therapy and/or other immunosuppressive therapy, as treatment for irAEs, for ≥ 14 days from Cycle 1, Day 1.
   3. Participants who experienced Grade 3 irAEs consisting of laboratory abnormalities that were asymptomatic and have now resolved to ≤ Grade 1 or baseline and participants who have been off steroid and/or other immunosuppressive therapy, as treatment for irAEs, for ≥ 30 days from Cycle 1, Day 1.
6. Concurrent malignancies are permitted if any one of the following applies:

   1. Previously treated malignancy for which all treatment of that malignancy was completed at least 2 years before enrollment and no evidence of disease exists, or
   2. With agreement from the Sponsor and Principal Investigator (PI), participants who have a concurrent malignancy that is clinically stable and does not require tumor-directed treatment are eligible to participate if the risk of the prior malignancy interfering with either safety or efficacy endpoints is very low, or
   3. With agreement from the Sponsor and PI, other malignancies may be permitted if the risk of the prior malignancy interfering with either safety or efficacy end points is very low.
7. Provide newly obtained core needle or incisional biopsy of a tumor lesion not previously irradiated. Fine needle aspiration is not acceptable.

   a. Biopsies should be obtained from sites that do not pose significant risk to the participant based on the tumor site and the procedure used. Biopsy sites/procedures including, but not limited to, the brain, open lung/mediastinum, pancreas, or endoscopic procedures extending beyond the esophagus, stomach, or bowel would be considered to pose a significant risk to the participant. Procedures to areas that are deemed by the Investigator to be of non-significant risk based on individual clinical scenarios will be permitted.
8. Measurable disease as defined by RECIST v1.1.

   a. Participants who do not have measurable disease by RECIST criteria but whose disease can be objectively measured through tumor markers or another disease specific standard are considered eligible.
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
10. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN).

    1. Participants who have liver lesions may be eligible if they have AST and ALT

       ≤ 3.0 x ULN.
    2. Participants with hepatocellular carcinoma (HCC) may be eligible provided they have AST and ALT that are ≤ 5.0 x ULN.
11. Hemoglobin ≥ 9 g/dL.
12. Total bilirubin ≤ 1.5 × ULN. Participants with liver lesions who do not have HCC and who have a total bilirubin < 2.0 x ULN may be eligible.

    1. Participants with HCC are eligible provided they have total bilirubin < 3.0 x ULN and are considered Child-Pugh Class A or Child-Pugh Class B7 (Child-Pugh Class B with a total Child-Pugh score not to exceed 7).
    2. Participants with Gilbert syndrome must have ≤ 3 x ULN and no liver lesions.
13. Creatinine clearance should be ≥ 30 mL/min as estimated by the Cockcroft-Gault equation.
14. Absolute neutrophil count ≥ 1.0 x 109/L.
15. Platelets count ≥ 75 x 109/L.
16. Participants must be capable of giving signed informed consent.
17. Evidence of stage IV prostate cancer (as defined by American Joint Committee of Cancer criteria) on previous bone, CT and/or MRI scan.
18. Ongoing androgen deprivation therapy (ADT) with a gonadotropin-releasing hormone (GnRH) analogue or a surgical/medical castration with testosterone level of ≤ 1.73 nmol/L (< 50 ng/dL).
19. Participants with skeletal system symptoms who are already on medications (eg, bisphosphonates and/or RANK ligand inhibitors) to strengthen bones are allowed if they were started ˃ 28 days before the first dose of study treatment.
20. Participants must have measurable disease per RECIST v 1.1.
21. Have received and progressed on prior secondary androgen receptor signaling inhibitor therapy (eg, abiraterone, enzalutamide, apalutamide).

Exclusion Criteria:

1. Participants who had a medical condition that required a surgical procedure and were subject to general anesthesia within 4 weeks prior to beginning protocol therapy are excluded except the use of general anesthesia during biopsy procedures, indicated for patient comfort and or safety will be permitted.
2. Pregnant or breastfeeding.
3. Significant gastrointestinal disorder(s) (eg, active Crohn disease or ulcerative colitis or a history of extensive gastric resection and/or small intestinal resection).
4. Has interstitial lung disease or active, noninfectious pneumonitis.
5. Has a transplanted organ or has undergone allogeneic bone marrow transplant.
6. Has received a live vaccine within 30 days prior to first dose.
7. Known hypersensitivity to a component of protocol therapy.

   a. Participants with known hypersensitivity to ipilimumab and/or nivolumab are excluded.
8. Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, clinically significant non-healing or healing wounds, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, significant pulmonary disease (shortness of breath at rest or on mild exertion), uncontrolled infection, or psychiatric illness/social situations that would limit compliance with study requirements.
9. Abnormal electrocardiograms (ECGs) that are clinically significant, clinically significant cardiac enlargement or hypertrophy, new bundle branch block or existing left bundle branch block, or signs of new, active ischemia.

   a. Participants with evidence of prior infarction who are New York Heart Association (NYHA) functional class II, III, or IV are excluded, as are participants with marked arrhythmia such as Wolff Parkinson White pattern or complete atrioventricular dissociation.*

   *Participants with complete or incomplete atrioventricular dissociation who have a pacemaker may be eligible for enrollment provided they are NYHA functional class I: "No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, or dyspnea (shortness of breath)."
10. Participants who experienced any ≥ Grade 3 symptomatic irAE on a prior immunotherapy study will be excluded from this study regardless of resolution of the irAE.
11. Any known, untreated, brain metastases. Treated participants must be stable 4 weeks after completion of treatment for brain metastases, and image-documented stability is required. Participants must have no clinical symptoms from brain metastases and have not required systemic corticosteroids > 10 mg/day prednisone or equivalent for ≥ 2 weeks prior to first dose of study intervention.
12. Has an active autoimmune disease requiring immunosuppression except for participants with isolated vitiligo, resolved childhood asthma or atopic dermatitis, controlled hypoadrenalism or hypopituitarism, and euthyroid participants with a history of Graves' disease.

    a. Participants with controlled hyperthyroidism must be negative for thyroglobulin and thyroid peroxidase antibodies and thyroid-stimulating immunoglobulin prior to study intervention administration.
13. Anticancer chemotherapy, radiotherapy, immunotherapy, or investigational agents within 14 days of first dose of study intervention, provided that all treatment-related AEs have resolved.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parker Institute for Cancer Immunotherapy, Study Director — Parker Institute for Cancer Immunotherapy
Locations (6):
- United States (6):
  - University of California, Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - M.D. Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ayers M, Lunceford J, Nebozhyn M, Murphy E, Loboda A, Kaufman DR, Albright A, Cheng JD, Kang SP, Shankaran V, Piha-Paul SA, Yearley J, Seiwert TY, Ribas A, McClanahan TK. IFN-gamma-related mRNA profile predicts clinical response to PD-1 blockade. J Clin Invest. 2017 Aug 1;127(8):2930-2940. doi: 10.1172/JCI91190. Epub 2017 Jun 26. PMID 28650338
- [Background] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- [Background] Chen PL, Roh W, Reuben A, Cooper ZA, Spencer CN, Prieto PA, Miller JP, Bassett RL, Gopalakrishnan V, Wani K, De Macedo MP, Austin-Breneman JL, Jiang H, Chang Q, Reddy SM, Chen WS, Tetzlaff MT, Broaddus RJ, Davies MA, Gershenwald JE, Haydu L, Lazar AJ, Patel SP, Hwu P, Hwu WJ, Diab A, Glitza IC, Woodman SE, Vence LM, Wistuba II, Amaria RN, Kwong LN, Prieto V, Davis RE, Ma W, Overwijk WW, Sharpe AH, Hu J, Futreal PA, Blando J, Sharma P, Allison JP, Chin L, Wargo JA. Analysis of Immune Signatures in Longitudinal Tumor Samples Yields Insight into Biomarkers of Response and Mechanisms of Resistance to Immune Checkpoint Blockade. Cancer Discov. 2016 Aug;6(8):827-37. doi: 10.1158/2159-8290.CD-15-1545. Epub 2016 Jun 14. PMID 27301722
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Feldmeyer L, Hudgens CW, Ray-Lyons G, Nagarajan P, Aung PP, Curry JL, Torres-Cabala CA, Mino B, Rodriguez-Canales J, Reuben A, Chen PL, Ko JS, Billings SD, Bassett RL, Wistuba II, Cooper ZA, Prieto VG, Wargo JA, Tetzlaff MT. Density, Distribution, and Composition of Immune Infiltrates Correlate with Survival in Merkel Cell Carcinoma. Clin Cancer Res. 2016 Nov 15;22(22):5553-5563. doi: 10.1158/1078-0432.CCR-16-0392. Epub 2016 May 10. PMID 27166398
- [Background] Gao J, Ward JF, Pettaway CA, Shi LZ, Subudhi SK, Vence LM, Zhao H, Chen J, Chen H, Efstathiou E, Troncoso P, Allison JP, Logothetis CJ, Wistuba II, Sepulveda MA, Sun J, Wargo J, Blando J, Sharma P. VISTA is an inhibitory immune checkpoint that is increased after ipilimumab therapy in patients with prostate cancer. Nat Med. 2017 May;23(5):551-555. doi: 10.1038/nm.4308. Epub 2017 Mar 27. PMID 28346412
- [Background] Gopalakrishnan V, Spencer CN, Nezi L, Reuben A, Andrews MC, Karpinets TV, Prieto PA, Vicente D, Hoffman K, Wei SC, Cogdill AP, Zhao L, Hudgens CW, Hutchinson DS, Manzo T, Petaccia de Macedo M, Cotechini T, Kumar T, Chen WS, Reddy SM, Szczepaniak Sloane R, Galloway-Pena J, Jiang H, Chen PL, Shpall EJ, Rezvani K, Alousi AM, Chemaly RF, Shelburne S, Vence LM, Okhuysen PC, Jensen VB, Swennes AG, McAllister F, Marcelo Riquelme Sanchez E, Zhang Y, Le Chatelier E, Zitvogel L, Pons N, Austin-Breneman JL, Haydu LE, Burton EM, Gardner JM, Sirmans E, Hu J, Lazar AJ, Tsujikawa T, Diab A, Tawbi H, Glitza IC, Hwu WJ, Patel SP, Woodman SE, Amaria RN, Davies MA, Gershenwald JE, Hwu P, Lee JE, Zhang J, Coussens LM, Cooper ZA, Futreal PA, Daniel CR, Ajami NJ, Petrosino JF, Tetzlaff MT, Sharma P, Allison JP, Jenq RR, Wargo JA. Gut microbiome modulates response to anti-PD-1 immunotherapy in melanoma patients. Science. 2018 Jan 5;359(6371):97-103. doi: 10.1126/science.aan4236. Epub 2017 Nov 2. PMID 29097493
- [Background] Haanen JBAG. Converting Cold into Hot Tumors by Combining Immunotherapies. Cell. 2017 Sep 7;170(6):1055-1056. doi: 10.1016/j.cell.2017.08.031. PMID 28886376
- [Background] Hegde PS, Karanikas V, Evers S. The Where, the When, and the How of Immune Monitoring for Cancer Immunotherapies in the Era of Checkpoint Inhibition. Clin Cancer Res. 2016 Apr 15;22(8):1865-74. doi: 10.1158/1078-0432.CCR-15-1507. PMID 27084740
- [Background] Herbst RS, Baas P, Kim DW, Felip E, Perez-Gracia JL, Han JY, Molina J, Kim JH, Arvis CD, Ahn MJ, Majem M, Fidler MJ, de Castro G Jr, Garrido M, Lubiniecki GM, Shentu Y, Im E, Dolled-Filhart M, Garon EB. Pembrolizumab versus docetaxel for previously treated, PD-L1-positive, advanced non-small-cell lung cancer (KEYNOTE-010): a randomised controlled trial. Lancet. 2016 Apr 9;387(10027):1540-1550. doi: 10.1016/S0140-6736(15)01281-7. Epub 2015 Dec 19. PMID 26712084
- [Background] Hodi FS, O'Day SJ, McDermott DF, Weber RW, Sosman JA, Haanen JB, Gonzalez R, Robert C, Schadendorf D, Hassel JC, Akerley W, van den Eertwegh AJ, Lutzky J, Lorigan P, Vaubel JM, Linette GP, Hogg D, Ottensmeier CH, Lebbe C, Peschel C, Quirt I, Clark JI, Wolchok JD, Weber JS, Tian J, Yellin MJ, Nichol GM, Hoos A, Urba WJ. Improved survival with ipilimumab in patients with metastatic melanoma. N Engl J Med. 2010 Aug 19;363(8):711-23. doi: 10.1056/NEJMoa1003466. Epub 2010 Jun 5. PMID 20525992
- [Background] Johnson DB, Estrada MV, Salgado R, Sanchez V, Doxie DB, Opalenik SR, Vilgelm AE, Feld E, Johnson AS, Greenplate AR, Sanders ME, Lovly CM, Frederick DT, Kelley MC, Richmond A, Irish JM, Shyr Y, Sullivan RJ, Puzanov I, Sosman JA, Balko JM. Melanoma-specific MHC-II expression represents a tumour-autonomous phenotype and predicts response to anti-PD-1/PD-L1 therapy. Nat Commun. 2016 Jan 29;7:10582. doi: 10.1038/ncomms10582. PMID 26822383
- [Background] Kvistborg P, Philips D, Kelderman S, Hageman L, Ottensmeier C, Joseph-Pietras D, Welters MJ, van der Burg S, Kapiteijn E, Michielin O, Romano E, Linnemann C, Speiser D, Blank C, Haanen JB, Schumacher TN. Anti-CTLA-4 therapy broadens the melanoma-reactive CD8+ T cell response. Sci Transl Med. 2014 Sep 17;6(254):254ra128. doi: 10.1126/scitranslmed.3008918. PMID 25232180
- [Background] Larkin J, Chiarion-Sileni V, Gonzalez R, Grob JJ, Cowey CL, Lao CD, Schadendorf D, Dummer R, Smylie M, Rutkowski P, Ferrucci PF, Hill A, Wagstaff J, Carlino MS, Haanen JB, Maio M, Marquez-Rodas I, McArthur GA, Ascierto PA, Long GV, Callahan MK, Postow MA, Grossmann K, Sznol M, Dreno B, Bastholt L, Yang A, Rollin LM, Horak C, Hodi FS, Wolchok JD. Combined Nivolumab and Ipilimumab or Monotherapy in Untreated Melanoma. N Engl J Med. 2015 Jul 2;373(1):23-34. doi: 10.1056/NEJMoa1504030. Epub 2015 May 31. PMID 26027431
- [Background] Maby P, Galon J, Latouche JB. Frameshift mutations, neoantigens and tumor-specific CD8(+) T cells in microsatellite unstable colorectal cancers. Oncoimmunology. 2015 Nov 24;5(5):e1115943. doi: 10.1080/2162402X.2015.1115943. eCollection 2016 May. PMID 27467916
- [Background] Maio M, Grob JJ, Aamdal S, Bondarenko I, Robert C, Thomas L, Garbe C, Chiarion-Sileni V, Testori A, Chen TT, Tschaika M, Wolchok JD. Five-year survival rates for treatment-naive patients with advanced melanoma who received ipilimumab plus dacarbazine in a phase III trial. J Clin Oncol. 2015 Apr 1;33(10):1191-6. doi: 10.1200/JCO.2014.56.6018. Epub 2015 Feb 23. PMID 25713437
- [Background] Momtaz P, Park V, Panageas KS, Postow MA, Callahan M, Wolchok JD, Chapman PB. Safety of Infusing Ipilimumab Over 30 Minutes. J Clin Oncol. 2015 Oct 20;33(30):3454-8. doi: 10.1200/JCO.2015.61.0030. Epub 2015 Jun 29. PMID 26124475
- [Background] Motzer RJ, Escudier B, McDermott DF, George S, Hammers HJ, Srinivas S, Tykodi SS, Sosman JA, Procopio G, Plimack ER, Castellano D, Choueiri TK, Gurney H, Donskov F, Bono P, Wagstaff J, Gauler TC, Ueda T, Tomita Y, Schutz FA, Kollmannsberger C, Larkin J, Ravaud A, Simon JS, Xu LA, Waxman IM, Sharma P; CheckMate 025 Investigators. Nivolumab versus Everolimus in Advanced Renal-Cell Carcinoma. N Engl J Med. 2015 Nov 5;373(19):1803-13. doi: 10.1056/NEJMoa1510665. Epub 2015 Sep 25. PMID 26406148
- [Background] Motzer RJ, Tannir NM, McDermott DF, Aren Frontera O, Melichar B, Choueiri TK, Plimack ER, Barthelemy P, Porta C, George S, Powles T, Donskov F, Neiman V, Kollmannsberger CK, Salman P, Gurney H, Hawkins R, Ravaud A, Grimm MO, Bracarda S, Barrios CH, Tomita Y, Castellano D, Rini BI, Chen AC, Mekan S, McHenry MB, Wind-Rotolo M, Doan J, Sharma P, Hammers HJ, Escudier B; CheckMate 214 Investigators. Nivolumab plus Ipilimumab versus Sunitinib in Advanced Renal-Cell Carcinoma. N Engl J Med. 2018 Apr 5;378(14):1277-1290. doi: 10.1056/NEJMoa1712126. Epub 2018 Mar 21. PMID 29562145
- [Background] Rizvi NA, Hellmann MD, Snyder A, Kvistborg P, Makarov V, Havel JJ, Lee W, Yuan J, Wong P, Ho TS, Miller ML, Rekhtman N, Moreira AL, Ibrahim F, Bruggeman C, Gasmi B, Zappasodi R, Maeda Y, Sander C, Garon EB, Merghoub T, Wolchok JD, Schumacher TN, Chan TA. Cancer immunology. Mutational landscape determines sensitivity to PD-1 blockade in non-small cell lung cancer. Science. 2015 Apr 3;348(6230):124-8. doi: 10.1126/science.aaa1348. Epub 2015 Mar 12. PMID 25765070
- [Background] Robert C, Schachter J, Long GV, Arance A, Grob JJ, Mortier L, Daud A, Carlino MS, McNeil C, Lotem M, Larkin J, Lorigan P, Neyns B, Blank CU, Hamid O, Mateus C, Shapira-Frommer R, Kosh M, Zhou H, Ibrahim N, Ebbinghaus S, Ribas A; KEYNOTE-006 investigators. Pembrolizumab versus Ipilimumab in Advanced Melanoma. N Engl J Med. 2015 Jun 25;372(26):2521-32. doi: 10.1056/NEJMoa1503093. Epub 2015 Apr 19. PMID 25891173
- [Background] Roy S, Trinchieri G. Microbiota: a key orchestrator of cancer therapy. Nat Rev Cancer. 2017 May;17(5):271-285. doi: 10.1038/nrc.2017.13. Epub 2017 Mar 17. PMID 28303904
- [Background] Schadendorf D, Hodi FS, Robert C, Weber JS, Margolin K, Hamid O, Patt D, Chen TT, Berman DM, Wolchok JD. Pooled Analysis of Long-Term Survival Data From Phase II and Phase III Trials of Ipilimumab in Unresectable or Metastatic Melanoma. J Clin Oncol. 2015 Jun 10;33(17):1889-94. doi: 10.1200/JCO.2014.56.2736. Epub 2015 Feb 9. PMID 25667295
- [Background] Thall PF, Simon RM, Estey EH. Bayesian sequential monitoring designs for single-arm clinical trials with multiple outcomes. Stat Med. 1995 Feb 28;14(4):357-79. doi: 10.1002/sim.4780140404. PMID 7746977
- [Background] Thompson ED, Zahurak M, Murphy A, Cornish T, Cuka N, Abdelfatah E, Yang S, Duncan M, Ahuja N, Taube JM, Anders RA, Kelly RJ. Patterns of PD-L1 expression and CD8 T cell infiltration in gastric adenocarcinomas and associated immune stroma. Gut. 2017 May;66(5):794-801. doi: 10.1136/gutjnl-2015-310839. Epub 2016 Jan 22. PMID 26801886
- [Background] Tumeh PC, Harview CL, Yearley JH, Shintaku IP, Taylor EJ, Robert L, Chmielowski B, Spasic M, Henry G, Ciobanu V, West AN, Carmona M, Kivork C, Seja E, Cherry G, Gutierrez AJ, Grogan TR, Mateus C, Tomasic G, Glaspy JA, Emerson RO, Robins H, Pierce RH, Elashoff DA, Robert C, Ribas A. PD-1 blockade induces responses by inhibiting adaptive immune resistance. Nature. 2014 Nov 27;515(7528):568-71. doi: 10.1038/nature13954. PMID 25428505
- [Background] Weber JS, D'Angelo SP, Minor D, Hodi FS, Gutzmer R, Neyns B, Hoeller C, Khushalani NI, Miller WH Jr, Lao CD, Linette GP, Thomas L, Lorigan P, Grossmann KF, Hassel JC, Maio M, Sznol M, Ascierto PA, Mohr P, Chmielowski B, Bryce A, Svane IM, Grob JJ, Krackhardt AM, Horak C, Lambert A, Yang AS, Larkin J. Nivolumab versus chemotherapy in patients with advanced melanoma who progressed after anti-CTLA-4 treatment (CheckMate 037): a randomised, controlled, open-label, phase 3 trial. Lancet Oncol. 2015 Apr;16(4):375-84. doi: 10.1016/S1470-2045(15)70076-8. Epub 2015 Mar 18. PMID 25795410
- [Background] Wolchok JD, Hoos A, O'Day S, Weber JS, Hamid O, Lebbe C, Maio M, Binder M, Bohnsack O, Nichol G, Humphrey R, Hodi FS. Guidelines for the evaluation of immune therapy activity in solid tumors: immune-related response criteria. Clin Cancer Res. 2009 Dec 1;15(23):7412-20. doi: 10.1158/1078-0432.CCR-09-1624. Epub 2009 Nov 24. PMID 19934295
- [Background] Wolchok JD, Chiarion-Sileni V, Gonzalez R, Rutkowski P, Grob JJ, Cowey CL, Lao CD, Wagstaff J, Schadendorf D, Ferrucci PF, Smylie M, Dummer R, Hill A, Hogg D, Haanen J, Carlino MS, Bechter O, Maio M, Marquez-Rodas I, Guidoboni M, McArthur G, Lebbe C, Ascierto PA, Long GV, Cebon J, Sosman J, Postow MA, Callahan MK, Walker D, Rollin L, Bhore R, Hodi FS, Larkin J. Overall Survival with Combined Nivolumab and Ipilimumab in Advanced Melanoma. N Engl J Med. 2017 Oct 5;377(14):1345-1356. doi: 10.1056/NEJMoa1709684. Epub 2017 Sep 11. PMID 28889792
- See also: Yervoy (ipilimumab) US Prescribing Information (USPI), April 2018 — https://packageinserts.bms.com/pi/pi_yervoy.pdf
- See also: Opdivo (nivolumab) US Prescribing Information (USPI), April 2018 — https://packageinserts.bms.com/pi/pi_opdivo.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- "Hot" Tumors for Advanced Metastatic Cancer: Participants with ≥ 15% CD8 cells in their tumor biopsies (ie, CD8 high tumors) will be treated with single-agent nivolumab. At the occurrence of disease progression (PD), participants will be allowed to add ipilimumab.
  Nivolumab Monotherapy: Single-agent nivolumab will be administered at 360 mg IV every 3 weeks (Q3W). Participants who continue to show clinical benefit after the first disease assessment will receive nivolumab 480 mg IV every 4 weeks (Q4W) until PD or intolerable toxicity.
Period: Overall Study
Arm/Group | "Hot" Tumors for Advanced Metastatic Cancer | "Cold" Tumors for Advanced Metastatic Cancer | "Hot" Tumors for Advanced Prostate Cancer | "Cold" Tumors for Advanced Prostate Cancer Cohort A | "Cold" Tumors for Advanced Prostate Cancer Cohort B
Started | 7 | 72 | 1 | 5 | 15
Completed | 1 | 13 | 1 | 1 | 8
Not Completed | 6 | 59 | 0 | 4 | 7
Not completed — Death | 4 | 37 | 0 | 2 | 6
Not completed — Lost to Follow-up | 1 | 5 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 15 | 0 | 0 | 1
Not completed — Patient medically unable to continue | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | "Hot" Tumors for Advanced Metastatic Cancer | "Cold" Tumors for Advanced Metastatic Cancer | "Hot" Tumors for Advanced Prostate Cancer | "Cold" Tumors for Advanced Prostate Cancer Cohort A | "Cold" Tumors for Advanced Prostate Cancer Cohort B | Total
Number analyzed (Participants) | 7 | 72 | 1 | 5 | 15 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 46 | 0 | 1 | 4 | 57
  >=65 years | 1 | 26 | 1 | 4 | 11 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 35 | 0 | 0 | 0 | 36
  Male | 6 | 37 | 1 | 5 | 15 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 9 | 0 | 0 | 0 | 9
  Not Hispanic or Latino | 7 | 63 | 1 | 5 | 15 | 91
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 5 | 0 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 7 | 0 | 1 | 1 | 9
  White | 6 | 45 | 1 | 3 | 14 | 69
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 15 | 0 | 1 | 0 | 17
Region of Enrollment [Number; unit: participants]
  United States | 7 | 72 | 1 | 5 | 15 | 100
Eastern Cooperative Oncology Group (ECOG) Performance Score [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) performance status is a widely-used scale to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine the appropriate treatment and prognosis.
  Here is a brief description of the ECOG performance status:
  * 0: Fully active, able to carry on all pre-disease performance without restriction.
  * 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework or office work. Population: Two participants did not have an ECOG performance score recorded at Screening and are excluded from analysis.
  Participants
    number analyzed (Participants) | 7 | 70 | 1 | 5 | 15 | 98
    0 | 4 | 23 | 0 | 0 | 4 | 31
    1 | 3 | 47 | 1 | 5 | 11 | 67
Primary Tumor Type [Count of Participants; unit: Participants] — The type of primary tumor diagnosed in the patient, as identified and reported by the investigator. This measure is derived from clinical assessments, imaging studies, histopathological evaluations, and/or medical records.
  Participants
    Prostate | 0 | 12 | 1 | 5 | 15 | 33
    Head and Neck | 3 | 6 | 0 | 0 | 0 | 9
    Colorectal | 0 | 7 | 0 | 0 | 0 | 7
    Sarcoma | 0 | 7 | 0 | 0 | 0 | 7
    Ovarian | 1 | 5 | 0 | 0 | 0 | 6
    Uterine | 0 | 4 | 0 | 0 | 0 | 4
    Breast | 0 | 3 | 0 | 0 | 0 | 3
    Hepatocellular cholangiocarcinoma | 0 | 3 | 0 | 0 | 0 | 3
    Neuroendocrine | 0 | 3 | 0 | 0 | 0 | 3
    Renal | 1 | 2 | 0 | 0 | 0 | 3
    Thyroid | 0 | 3 | 0 | 0 | 0 | 3
    Urethral | 1 | 0 | 0 | 0 | 0 | 1
    Gastroesophageal | 1 | 0 | 0 | 0 | 0 | 1
    Cervix | 0 | 2 | 0 | 0 | 0 | 2
    Gastric | 0 | 2 | 0 | 0 | 0 | 2
    Non-small cell lung | 0 | 2 | 0 | 0 | 0 | 2
    Pancreatic | 0 | 2 | 0 | 0 | 0 | 2
    Pelvic | 0 | 2 | 0 | 0 | 0 | 2
    Peritoneal | 0 | 2 | 0 | 0 | 0 | 2
    Hepatocellular carcinoma | 0 | 1 | 0 | 0 | 0 | 1
    Merkel cell | 0 | 1 | 0 | 0 | 0 | 1
    Penile | 0 | 1 | 0 | 0 | 0 | 1
    Retroperitoneal teratoma | 0 | 1 | 0 | 0 | 0 | 1
    Papilla of vater | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CBR) of Nivolumab With or Without Ipilimumab
Description: CBR is defined as the percentage of participants who show clinical benefit, defined as obtaining a complete response (CR; disappearance of all target and non-target lesions), partial response (PR; ≥ 30% decrease in the sum of the longest diameter of target lesions), or stable disease (SD) for ≥ 6 months, as determined by Response Evaluation Criteria in Solid Tumours (RECIST) v1.1.
Time Frame: Initiation of study drug through radiographic progression or initiation of new anti-cancer therapy, whichever occurred first, up to 43 months
Measure: Count of Participants; unit: Participants
Arm/Group | "Hot" Tumors for Advanced Metastatic Cancer | "Cold" Tumors for Advanced Metastatic Cancer | "Hot" Tumors for Advanced Prostate Cancer | "Cold" Tumors for Advanced Prostate Cancer Cohort A | "Cold" Tumors for Advanced Prostate Cancer Cohort B
Number analyzed (Participants) | 7 | 72 | 1 | 5 | 15
Participants | 1 | 18 | 1 | 1 | 3

2. Primary Outcome: Percentage of Participants Whose Tumors Convert From CD8 Low (<15% Tumoral CD8) to CD8 High (>=15%).
Description: Percentage of participants in the nivolumab plus ipilimumab ("CD8 low") arm whose tumors convert from CD8 low (<15%) to CD8 high (>=15%) as measured by the percentage of tumoral CD8 cells. Participants in the CD8 high arms are not evaluated for this outcome.
  On-treatment biopsies for the advanced metastatic cancer cohort were scheduled for as early as possible after the 2nd and 4th doses of ipilimumab (Day 2 - 10 of Cycle 2 and Cycle 6, respectively). On-treatment biopsies for the advanced prostate cancer cohort were scheduled for within 3 days (+/-) of the 2nd and 4th doses of nivolumab (Day 22 of Cycle 1 and Cycle 2, respectively).
Time Frame: From initiation of study intervention through the 2nd on-treatment tumor biopsy, up to 8 months
Population: Only CD8 low participants with an on-treatment biopsy are included in the analysis population for this outcome. Participants in the CD8 high arms and participants without an on-treatment biopsy are not evaluated for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | "Cold" Tumors for Advanced Metastatic Cancer | "Cold" Tumors for Advanced Prostate Cancer Cohort A | "Cold" Tumors for Advanced Prostate Cancer Cohort B
Number analyzed (Participants) | 39 | 3 | 8
Participants | 14 | 1 | 1

3. Secondary Outcome: Number of Participants With Treatment-related Adverse Events (TRAE)
Description: Investigators recorded adverse events (AEs) during each participant encounter. AE severity was assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, which grades AEs on a 1 to 5 scale: Grades 1 and 2 indicate mild to moderate events; Grade 3 denotes severe events; Grades 4 and 5 signify life-threatening or fatal outcomes.
  A TRAE is defined as any event that either occurs after the initiation of study intervention, having been absent at baseline, or, if present at baseline, appears to have worsened in severity or frequency, that is deemed 'Possibly', 'Probably', or 'Definitely' related to the intervention by the Investigator.
  All TRAEs were collected from the time the participant signed informed consent until 100 days after the last dose of study intervention. Prior to initiation of study intervention, only TRAEs that were related to a protocol mandated intervention, including those that occurred prior to being assigned to a study arm, were reported.
Time Frame: From signing informed consent (prior to Screening) through 100 days after last dose, up to 43 months.
Measure: Count of Participants; unit: Participants
Arm/Group | "Hot" Tumors for Advanced Metastatic Cancer | "Cold" Tumors for Advanced Metastatic Cancer | "Hot" Tumors for Advanced Prostate Cancer | "Cold" Tumors for Advanced Prostate Cancer Cohort A | "Cold" Tumors for Advanced Prostate Cancer Cohort B
Number analyzed (Participants) | 7 | 72 | 1 | 5 | 15
Participants
  Any Treatment-related adverse event (TRAE) | 4 | 58 | 1 | 4 | 12
  Grade 3 or Grade 4 TRAE | 0 | 20 | 0 | 2 | 6
  Grade 5 TRAE | 0 | 0 | 0 | 0 | 0
  Serious TRAE | 0 | 10 | 0 | 1 | 6
  TRAE leading to treatment discontinuation | 0 | 4 | 0 | 0 | 5

4. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate (ORR) is defined as the percentage of participants who attain a best overall response of complete response (CR; disappearance of all target and non-target lesions) or partial response (PR; >= 30% decrease in the sum of the longest diameter of target lesions), as determined by Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | "Hot" Tumors for Advanced Metastatic Cancer | "Cold" Tumors for Advanced Metastatic Cancer | "Hot" Tumors for Advanced Prostate Cancer | "Cold" Tumors for Advanced Prostate Cancer Cohort A | "Cold" Tumors for Advanced Prostate Cancer Cohort B
Number analyzed (Participants) | 7 | 72 | 1 | 5 | 15
Participants | 1 | 14 | 0 | 0 | 1

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from initiation of study intervention to the date of first documented radiographic progression of disease or date of death due to any cause, whichever occurred first. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Initiation of study drug through death, radiographic progression or initiation of new anti-cancer therapy, whichever occurred first, up to 43 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | "Hot" Tumors for Advanced Metastatic Cancer | "Cold" Tumors for Advanced Metastatic Cancer | "Hot" Tumors for Advanced Prostate Cancer | "Cold" Tumors for Advanced Prostate Cancer Cohort A | "Cold" Tumors for Advanced Prostate Cancer Cohort B
Number analyzed (Participants) | 7 | 72 | 1 | 5 | 15
months | 2.0 [1.1 to NA] — Upper confidence limit is not estimable due to insufficient number of participants with events. | 2.3 [2.0 to 4.3] | NA [NA to NA] — Median and confidence limits are not estimable due to insufficient number of participants with events. | 3.7 [1.1 to NA] — Upper confidence limit is not estimable due to insufficient number of participants with events. | 5.7 [2.0 to 7.9]

6. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from initiation of study intervention until death due to any cause. Participants not reported as having died at the time of analysis were censored at the most recent contact date they were known to be alive.
Time Frame: From initiation of study drug until death due to any cause, up to 43 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | "Hot" Tumors for Advanced Metastatic Cancer | "Cold" Tumors for Advanced Metastatic Cancer | "Hot" Tumors for Advanced Prostate Cancer | "Cold" Tumors for Advanced Prostate Cancer Cohort A | "Cold" Tumors for Advanced Prostate Cancer Cohort B
Number analyzed (Participants) | 7 | 72 | 1 | 5 | 15
months | 15.8 [12.1 to NA] — Upper confidence limit is not estimable due to insufficient number of participants with events. | 13.9 [8.9 to 21.1] | NA [NA to NA] — Median and confidence limits are not estimable due to insufficient number of participants with events. | NA [1.1 to NA] — Median and confidence limits are not estimable due to insufficient number of participants with events. | NA [4.9 to NA] — Median and confidence limits are not estimable due to insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: From initiation of study drug until death due to any cause, up to 43 months. All adverse events (AEs), regardless of relationship to study drug, were collected from the time the participant signed informed consent until 100 days after the last dose of study intervention. Serious Adverse Events (SAEs) that occurred after the end of the AE reporting period (100-days post last dose) and that were considered to be reasonably related to the study drug by the investigator, were also collected.
Description: Investigators recorded AEs during each participant encounter. All AEs, regardless of relationship to study drug, were collected from the time the participant signed informed consent until 100 days after the last dose of study intervention. Prior to initiation of study intervention, only AEs that were related to a protocol mandated intervention (e.g. biopsy), including those that occurred prior to being assigned to a study arm, were collected.
Arm/Group | "Hot" Tumors for Advanced Metastatic Cancer | "Cold" Tumors for Advanced Metastatic Cancer | "Hot" Tumors for Advanced Prostate Cancer | "Cold" Tumors for Advanced Prostate Cancer Cohort A | "Cold" Tumors for Advanced Prostate Cancer Cohort B
All-Cause Mortality (participants affected / at risk) | 4/7 | 39/72 | 0/1 | 2/5 | 6/15
Serious Adverse Events (participants affected / at risk) | 2/7 | 30/72 | 0/1 | 2/5 | 8/15
Other Adverse Events (participants affected / at risk) | 7/7 | 71/72 | 1/1 | 5/5 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | "Hot" Tumors for Advanced Metastatic Cancer (N=7) | "Cold" Tumors for Advanced Metastatic Cancer (N=72) | "Hot" Tumors for Advanced Prostate Cancer (N=1) | "Cold" Tumors for Advanced Prostate Cancer Cohort A (N=5) | "Cold" Tumors for Advanced Prostate Cancer Cohort B (N=15)
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Hypophysitis (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Thyroiditis (Endocrine disorders) | 0 | 2 | 0 | 0 | 0
Retinal vascular disorder (Eye disorders) | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 4 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 1
Amylase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 2 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Immune-Mediated Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Adrenocortical Insufficiency Acute (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Immune-Mediated Adrenal Insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Immune-Mediated Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Covid-19 Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood Bilirubin Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Guillain-Barre Syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Medical Device Site Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | "Hot" Tumors for Advanced Metastatic Cancer (N=7) | "Cold" Tumors for Advanced Metastatic Cancer (N=72) | "Hot" Tumors for Advanced Prostate Cancer (N=1) | "Cold" Tumors for Advanced Prostate Cancer Cohort A (N=5) | "Cold" Tumors for Advanced Prostate Cancer Cohort B (N=15)
Alanine Aminotransferase Increased (Investigations) | 0 | 6 | 0 | 1 | 3
Amylase Increased (Investigations) | 0 | 2 | 0 | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 9 | 0 | 1 | 3
Blood Creatinine Increased (Investigations) | 1 | 10 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 4 | 0 | 0 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 1 | 1 | 0 | 1 | 0
Blood Thyroid Stimulating Hormone Increased (Investigations) | 0 | 4 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 11 | 0 | 0 | 0
Low Density Lipoprotein Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 5 | 0 | 0 | 0
Pancreatic Enzymes Increased (Investigations) | 0 | 0 | 0 | 0 | 2
Sars-Cov-2 Test Positive (Investigations) | 0 | 0 | 0 | 1 | 0
Thyroid Function Test Abnormal (Investigations) | 0 | 0 | 0 | 0 | 1
Thyroxine Decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 1 | 0 | 0 | 0 | 0
Tri-Iodothyronine Decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Troponin I Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Troponin Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Weight Decreased (Investigations) | 1 | 5 | 0 | 0 | 4
Weight Increased (Investigations) | 0 | 0 | 0 | 0 | 1
White Blood Cell Count Decreased (Investigations) | 1 | 1 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 12 | 0 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 13 | 0 | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 21 | 0 | 1 | 3
Dry Mouth (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 18 | 0 | 1 | 5
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 6 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 13 | 0 | 1 | 4
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 13 | 0 | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 7 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 4 | 0 | 2 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 8 | 0 | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 6 | 0 | 0 | 1
Facial pain (General disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 36 | 1 | 3 | 4
Influenza like illness (General disorders) | 0 | 4 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 4 | 1 | 1 | 0
Pyrexia (General disorders) | 1 | 7 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 10 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 11 | 0 | 0 | 3
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 6 | 0 | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 12 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 0 | 2
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Dermatitis Bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 12 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 15 | 1 | 2 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 6 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Body tinea (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Campylobacter Colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Coronavirus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Oral Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Otitis Externa (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Penile Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 3 | 0 | 0 | 1
Skin Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 4 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 3 | 0 | 1 | 1
Adrenal Insufficiency (Endocrine disorders) | 0 | 3 | 0 | 1 | 2
Hyperthyroidism (Endocrine disorders) | 1 | 3 | 0 | 1 | 2
Hypophysitis (Endocrine disorders) | 1 | 1 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 2 | 8 | 0 | 0 | 3
Thyroiditis (Endocrine disorders) | 0 | 1 | 0 | 1 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 13 | 0 | 0 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 18 | 0 | 1 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Cystitis Noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 14 | 0 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 3 | 0 | 1 | 2
Insomnia (Psychiatric disorders) | 0 | 7 | 0 | 0 | 2
Bell's Palsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 6 | 0 | 0 | 0
Haemorrhage Intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 11 | 0 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Sinus Node Dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 0 | 0 | 1
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Extradural Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 0 | 0 | 0
Embolism Venous (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 7 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 3 | 0 | 1 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 1 | 2 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Abscess drainage (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Trial Site and/or Co-Principal Investigators may publish or present Study Data and other results of the Study from the Trial Site individually upon the first to occur of: (i) twelve (12) months after conclusion, abandonment, or termination of the Study at all Affiliated Research Institutions, or (ii) after Parker Institute for Cancer Immunotherapy (PICI) confirms in writing there will not be a multi-site Study publication.

DOCUMENTS (2):
  • Study Protocol (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT03651271/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT03651271/SAP_001.pdf